CLINICAL TRIAL: NCT03236142
Title: The Single Anastomosis, 300 cm Loop, Duodenal Switch (SIPS) Results in Less Nutritional Deficiencies Than the Standard Duodenal Switch (DS) Operation: A Multicenter, Randomized Controlled Trial
Brief Title: DS vs SIPS-Bariatric Surgery Comparasion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reading Health System (Other)
Responsible Party: Principal Investigator, Stephan Myers, MD, Stephan Myers, MD, FACS, Medical Director, Principal Investigator, Reading Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB 016-16
Record Dates: First submitted 2017-06-30; First posted 2017-08-01 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Bariatric Surgery Candidate
Keywords: bariatric; duodenal switch; DS; weight loss surgery; SIPS; Single Anastomosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Duodenal Switch (DS) (Active Comparator)
  Interventions: Procedure: Standard Duodenal Switch Operation
- Single Anastomosis, 300 cm Loop, Duodenal Switch (SIPS) (Experimental)
  Interventions: Procedure: SIPS Operation

INTERVENTIONS:
Procedure: SIPS Operation — The SIPS modification of the DS operation entails one less division of the small intestine and one less anastomosis, thereby reducing the time of the procedure.
  Arms: Single Anastomosis, 300 cm Loop, Duodenal Switch (SIPS)
Procedure: Standard Duodenal Switch Operation
  Arms: Standard Duodenal Switch (DS)

SUMMARY:
The aim of this study is to answer the question of whether the single anastomosis, 300 cm loop, duodenal switch (SIPS) is an equally effective, safe, simpler operation with less nutritional and surgical risks than the standard duodenal switch (DS) operation. Please note, this study does not provide a stipend or coverage for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 40 to 65
* Agree to not use weight loss medications for the length of the study
* Compliance with standards of surgical program

Exclusion Criteria:

* Patients with a history of previous bariatric surgery except for patients who have had a previous gastric sleeve
* Previous complex abdominal surgery
* Poorly controlled medical or psychiatric disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Vitamin A Deficiency | 36 months post surgery
  Proportion of patients with a vitamin A deficiency

SECONDARY OUTCOMES:
Vitamin D, zinc, copper, and albumin | 36 months post surgery
  Proportion of patients with vitamin D, zinc, copper, and albumin deficiency
Frequency of stools | 36 months post surgery
  Amount of stools per day
Length of Operation | Date of operation
  Length of surgical procedure in time
Percentage of excess weight lost | 36 months post surgery
  Weight in excess of a body mass index (BMI) of 25.0 lost
Body Mass Index (BMI) | 36 months post surgery
  Body mass index (weight in kilograms divided by height in meters squared

CONTACTS AND LOCATIONS:
Locations (1):
- Reading Health Physician Network Weight Management Center, West Reading, Pennsylvania, United States